CLINICAL TRIAL: NCT05069233
Title: Feasibility of the Magnetically Controlled Capsule Endoscopy in One Time Visualization of the Upper Gastrointestinal Tract and Small Intestine
Brief Title: Magnetically Controlled Capsule Endoscopy in Visualization of the UGI and Small Intestine
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Collaborators: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Zhuan Liao, Professor, Changhai Hospital
Other Study IDs: MCE for UGI+SB
Record Dates: First submitted 2021-09-17; First posted 2021-10-06 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Stomach Diseases; Small Intestine Disease
Keywords: capsule endoscopy
MeSH Terms: conditions — Stomach Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- UGI+SB: Patients who underwent combined upper digestive tract and small intestine examination under MCE.
  Interventions: Other: UGI+SB

INTERVENTIONS:
Other: UGI+SB — Patients who underwent combined upper digestive tract and small intestine examination under MCE.

SUMMARY:
In this study, we retrospectively analyzed the videos of combined upper digestive tract and small intestine examination under MCE, so as to clarify the feasibility and diagnostic efficacy of MCE in one-time examination of the upper gastrointestinal and small intestinal mucosa.

DETAILED DESCRIPTION:
Magnetically controlled capsule endoscopy (MCE), with equally favorable diagnostic accuracy as conventional endoscopy, has become a painless noninvasive diagnostic modality in clinical practice. The more than 8 hours battery life of the MCE enables a further examination of the small bowel. In addition, it has been demonstrated that magnetic steering of capsule endoscopy improves the completion rate of small bowel examination by facilitating passage of the capsule through the pylorus, which further supported MCE as a practical modality for examination of both the stomach and small bowel. In this study, we retrospectively analyzed the videos of combined upper digestive tract and small intestine examination under MCE, so as to clarify the feasibility and diagnostic efficacy of MCE in one-time examination of the upper gastrointestinal and small intestinal mucosa.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old.
2. Those who underwent upper gastrointestinal and small intestinal mucosal examination under magnetically controlled capsule endoscopy at Shanghai Changhai Hospital and Chinese PLA General Hospital after January 2020.
3. Able to provide informed consent.

Exclusion Criteria:

1. Patients who fail to follow the prescribed procedures for magnetically controlled capsule endoscopy;
2. Patients who only undergo gastric examination under magnetically controlled capsule endoscopy;
3. Patients who only undergo small bowel examination under magnetic control capsule endoscopy;
4. The patient's basic information in the database is incomplete；
5. Patient fail to be followed up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who underwent upper gastrointestinal and small intestinal mucosal examination under MCE at Shanghai Changhai Hospital and Chinese PLA General Hospital after January 2020.
Sampling Method: Probability Sample
Enrollment: 593 (Estimated)
Dates: Start 2021-09-27 (Actual); Primary Completion 2021-12-28 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Success rate of UGI and small-bowel examination | 2 weeks
  The success rate of upper gastrointestinal tract and small-bowel examination under MCE is evaluated by the technical success rate, a composite outcome including the successful viewing of esophagus, stomach and duodenum, and complete small-bowel examination.

SECONDARY OUTCOMES:
Visualization of the esophagus | 2 weeks
  Visualization of the esophagus indicated by the number of images captured for Z-line and how many quadrants of the Z-line were observed. Circumferential visualization of the Z-line is defined by quadrants as follows: less than 2 quadrants (< 50%) observed; at least 2 quadrants (50%-75%) observed; at least 3 quadrants (>75%) observed; and entire structure (100%) observed.
Visualization score of the gastric mucosa | 2 weeks
  Visualization score of the gastric mucosa To objectively evaluate the complete visualization of the gastric mucosa in the 6 anatomic landmarks (cardia, fundus, body, angulus, antrum, and pylorus), a 3-point grading scale was used: 1, poor (<70% of the mucosa was observed), 2, fair (70%-90% of the mucosa was observed), and 3, good (>90% of the mucosa was observed).
Visualization of the small bowel | 2 weeks
  Visualization of the small bowel was determined by the percentage of time during which the small-bowel view was clear, defined as not obscured more than 50% of the screen view. The clear-viewing percentage of the total small-bowel transit time assessed by a 4-point scale :0, less than 25%; 1, 25% to 49%; 2, 50% to 75%; and 3, greater than 75%.
Examination time of esophagus, stomach, duodenum and small bowel | 1 month
  Examination-related parameters included esophageal transit time (ETT), gastric examination time (GET), gastric transit time (GTT), pylorus transit time (PTT), small bowel transit time (SBTT). ETT is defined as the time between the first esophageal image and the first gastric image. GTT is defined as the time between the first gastric image and the first duodenal image. GET is defined as the time for examination of gastric primary anatomic landmarks twice. PTT is defined as the time between the first pyloric image and the first duodenal image. SBTT is defined as the time between the first duodenal image and the first cecal image.
Detection rate of lesions | 1 month
  The detection rate of lesions in different digestive part (esophagus, stomach, duodenum, small intestine) found by MCE.
Adverse events during MCE procedure | 1 month
  The presence of any adverse events during MCE procedure will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Zhuan Liao, Principal Investigator — Changhai Hospital,Shanghai,China
Locations (1):
- Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liao Z, Hou X, Lin-Hu EQ, Sheng JQ, Ge ZZ, Jiang B, Hou XH, Liu JY, Li Z, Huang QY, Zhao XJ, Li N, Gao YJ, Zhang Y, Zhou JQ, Wang XY, Liu J, Xie XP, Yang CM, Liu HL, Sun XT, Zou WB, Li ZS. Accuracy of Magnetically Controlled Capsule Endoscopy, Compared With Conventional Gastroscopy, in Detection of Gastric Diseases. Clin Gastroenterol Hepatol. 2016 Sep;14(9):1266-1273.e1. doi: 10.1016/j.cgh.2016.05.013. Epub 2016 May 20. PMID 27211503
- [Background] Jiang X, Qian YY, Liu X, Pan J, Zou WB, Zhou W, Luo YY, Chen YZ, Li ZS, Liao Z. Impact of magnetic steering on gastric transit time of a capsule endoscopy (with video). Gastrointest Endosc. 2018 Oct;88(4):746-754. doi: 10.1016/j.gie.2018.06.031. Epub 2018 Jul 11. PMID 30005825
- [Background] Luo YY, Pan J, Chen YZ, Jiang X, Zou WB, Qian YY, Zhou W, Liu X, Li ZS, Liao Z. Magnetic Steering of Capsule Endoscopy Improves Small Bowel Capsule Endoscopy Completion Rate. Dig Dis Sci. 2019 Jul;64(7):1908-1915. doi: 10.1007/s10620-019-5479-z. Epub 2019 Feb 6. PMID 30725289
- [Background] Chen X, Gao F, Zhang J. Screening for Gastric and Small Intestinal Mucosal Injury with Magnetically Controlled Capsule Endoscopy in Asymptomatic Patients Taking Enteric-Coated Aspirin. Gastroenterol Res Pract. 2018 Nov 15;2018:2524698. doi: 10.1155/2018/2524698. eCollection 2018. PMID 30581462
- [Derived] Liu YW, Wang YC, Zhu JH, Jiang X, Zhou W, Zhang J, Liao Z, Linghu EQ. Magnetically controlled capsule endoscopy in one-time gastro-small intestinal joint examination: a two-centre experience. BMC Gastroenterol. 2022 May 4;22(1):222. doi: 10.1186/s12876-022-02302-0. PMID 35509022